CLINICAL TRIAL: NCT05232643
Title: A Multicenter Prospective Observational Double Cohort Study to Evaluate the Associations Between Clinical Characteristics and Use of Oral Anticoagulants in Italian Elderly Patients Suffering From NVAF.
Brief Title: A Study Evaluating the Associations Between Clinical Characteristics and Use of Oral Anticoagulants in Italian Elderly Participants With Non-Valvular Atrial Fibrillation
Acronym: PRESBUS
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-754
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non-Valvular Atrial Fibrillation (NVAF)
Keywords: Atrial fibrillation; Oral Anticoagulants
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Cohort 1: Non-valvular atrial fibrillation (NVAF) participants administered oral anticoagulants (OAs)
- Cohort 2: Non-valvular atrial fibrillation (NVAF) participants not administered oral anticoagulants

SUMMARY:
The purpose of this study is to provide real-world data useful to address the factors associated to the administration of oral anticoagulants in the elderly population affected by non-valvular atrial fibrillation (NVAF), in Italy, and it's persistence rate after one year.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Diagnosis of any type (e.g. persistent, permanent, paroxysmal) of Non-Valvular Atrial Fibrillation (NVAF) documented in the participant's medical chart based on electrocardiogram (ECG) results, or diagnosed at enrollment
* Naïve to anticoagulant treatments, or not having received anticoagulant treatments during the 6 months prior to enrollment
* Multidimensional geriatric assessment (MGA) performed at enrollment, or anyway no more than 3 months before in case of stable disease (i.e. no relevant events) in the previous 3 months

Exclusion Criteria:

* Valvular atrial fibrillation (AF) due to artificial heart valve
* Medical conditions (apart from NVAF) requiring anticoagulant therapy (such as deep vein thrombosis or pulmonary embolism)
* Use of inappropriate direct-acting oral anticoagulant (DOAC) doses based on the current summary of product characteristics (SmPC) for any drugs

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study target population will be composed of elderly participants with diagnosis of Non-valvular atrial fibrillation (NVAF), managed in Italian geriatric departments/clinics.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Anticoagulant (OA) cohort: Distribution of participants starting any type of anticoagulant direct-acting oral anticoagulant (DOAC) or Vitamin K antagonist (VKA) treatment | At Enrollment, up to 12 months
Non-Anticoagulant (Not-OA) cohort: Distribution of participants not starting any type of anticoagulant (DOAC) or (VKA) treatment | At Enrollment, up to 12 months
Treatment switch: Change of antithrombotic drug (in terms of active principle) during the 12-month observational period | Up to approximately 12 months
Distribution of participants with persistence to the first treatment strategy: No switches nor interruptions of greater than 60 days in the first administered antithrombotic strategy (including no treatments) during the 12-month observational period | Up to approximately 12 months
Distribution of participants with net clinical outcomes defined as occurrence of stroke, systemic embolism, major bleeding or death | Up to approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Milan, MI, Italy

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm